CLINICAL TRIAL: NCT05551988
Title: Predictors of Foot Amputation in Diabetic Foot Ulcers; A Retrospective Study From Pakistan
Brief Title: Predictors of Foot Amputation in Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Bolan Medical Complex Hospital Quetta Pakistan (Other)
Responsible Party: Principal Investigator, Taimoor Hussain, Medical Officer, Bolan Medical Complex Hospital Quetta Pakistan
Other Study IDs: BUMHS/IRB/22
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Foot; Amputation; Antibiotic Resistant Strain; Diabetic Foot Ulcer
Keywords: antimicrobial resistance; antibiotic resistance; risk factors of amputation; predictors of amputation
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- diabetic foot ulcer patients: Diabetic foot ulcer patients with and without diabetic foot amputation
  Interventions: Other: Retrospective observational study of diabetic foot ulcer

INTERVENTIONS:
Other: Retrospective observational study of diabetic foot ulcer — This is a retrospective observational study of antibiotic resistance and risk factors of amputation in diabetic foot ulcer patients

SUMMARY:
Diabetes affects 463 million population of the world. Diabetic foot is one of the complications of uncontrolled diabetes which can lead to amputation in 5- 24% of non-healing diabetic foot ulcers. Every 30 seconds a lower extremity is amputated in the world due to diabetes.

This is a retrospective study conducted in Balochistan, Pakistan. In this study investigators explored the risk factor of amputation in diabetic patients. Baseline characteristics, clinical profile, and lab tests were retrieved retrospectively and presented in the forms of tables. Investigators compared the categorical variables in amputees vs non-amputees and analyzed associated risk factors of amputation.

DETAILED DESCRIPTION:
Proposal

In 2019 around 463 million (9.3%) of the global adult population (20-79 years) were estimated to be living with diabetes. This is a 62% increase from 2009 prevalence data which is projected to increase by another 10.9% (700 million) by 2045. What is surprising and more concerning is that almost half of the affected do not know they have diabetes. Pakistan with 19.6 million diabetics ranks fourth in terms of prevalence.

Uncontrolled diabetes leads to grave complications like diabetic retinopathy, neuropathy, nephropathy, and cardiovascular complications. Diabetic foot is one of the complications that causes significant disability. The global diabetic foot ulcer prevalence was 6.3% - 5.5% in Asia and with 13% in north America (13%). Although, majority (60-80%) of foot ulcers will heal, 5-24% of the remaining active ulcers will in the long run cause limb amputation within 6 to 18 months after the first evaluation. In fact, every 30 seconds in the world, a lower limb is amputated due to diabetes.

Diabetic foot amputations are associated with several risk factors, including peripheral vascular disease (PVD), neuropathy, longer diabetes duration, nephropathy, older age, poor glycemic control, comorbidities like coronary artery disease (CAD), preventive foot care, socioeconomic status, male gender, smoking, hypertension, and hyperlipidemia. Diabetic wound care management and foot care awareness and habits also play a definitive role in the outcome.

In this study investigators explored the baseline demographic, clinical, and lab investigations profile of diabetic foot patients visiting tertiary care hospitals of Baluchistan, Pakistan. Investigators also explored the associated risk factors of amputations in patients. The regional epidemiological knowledge and identifying the risk factors will guide physicians to improve patients' quality of life and reduce the economic burden for both the patient and the health care system.

Rationale of the study:

Antimicrobial surveillance studies of diabetic foot are the need of time to detect any variations in regional microbiological profile and rise in antimicrobial resistance, before it turns into a major public health nightmare. Addressing the risk factors of amputation in diabetic foot ulcer patients can avoid this dreadful complication. In this study investigators have attempted to address this void in regional data of diabetic foot. The results of this study will also guide physicians regarding appropriate choice of antibiotics, discourage indiscriminate abuse of antibiotics both by physicians and public, encourage practice of culture studies based treatment.

Operational definitions:

Diabetes Mellitus: Diagnosed at an HbA1C of greater than or equal to 6.5%; or a fasting blood glucose of more 126 mg/dl or higher Diabetic foot: Defined as a foot affected by ulceration that is associated with neuropathy and/or peripheral arterial disease of the lower limb in a patient with diabetes.

Hypertension: Previous medication of anti-hypertensive drug or a BP ≥ 140/90 mmHg).

Antibiotic resistance happens when germs like bacteria and fungi develop the ability to defeat the drugs designed to kill them. That means the germs are not killed and continue to grow.

Antibiotic resistance: When germs like bacteria and fungi develop the ability to defeat the drugs designed to kill them. That means the germs are not killed and continue to grow.

Multidrug resistance (MDR): Defined as acquired non-susceptibility to at least one agent in three or more antimicrobial categories, Extremely drug resistance (XDR): Defined as non-susceptibility to at least one agent in all but two or fewer antimicrobial categories (i.e. bacterial isolates remain susceptible to only one or two categories) Pan Drug resistance (PDR): Defined as non-susceptibility to all agents in all antimicrobial categories.

Duration and size of ulcer: Calculated by multiplying longest and widest diameters and expressed in centimeter square. Ulcers were graded using Wagner classification system, grade I (superficial ulcer or ulcer of subcutaneous tissue), grade II (ulcers extended into tendon, bone, or capsule), grade III (deep ulcer with osteomyelitis, or abscess), and grade IV (gangrene of toes). Subjects with grade 0 (uninfected lesions/ intact skin/ healed ulcers) were debarred from the study.

Amputation: Defined as the complete loss in the transverse anatomical plane of any part of the lower limb.

Diagnosis of infection involving bone: Done by either using a sterile probe in exposed bone or evidence obtained from plain radiographs.

Data collection procedure: Baseline characteristics of patients such as age, gender, residence district, rural or urban, education, income, HbA1c level, presence or absence of; neuropathy, peripheral arterial disease, amputation, grade and location of ulcer, and comorbidities will be retrieved from records and patient files. Incase of missing data patients shall be contacted for any previous records as needed.

Statistical analysis:

Quantitative variables represented as means ± standard deviation and categorical data as a percentage (%). SPSS and Microsoft Excel will be used to analyze the data . Chi square will be used to analyze for any difference between amputees and non amputees. Univariate logistic regression analysis will be applied to determine the odds ratio of variables as risk factors in amputees vs non amputees. Significant variable in univariate analysis will be entered in to multivariate logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic foot patients (male and female) aged 18 and above;
* Patients visiting Endocrine department of tertiary care hospitals of Balochistan, Pakistan

Exclusion Criteria:

* Patients who have received prior treatment with antibiotics in the last one month
* Patient with end stage renal disease requiring regular hemodialysis
* Those with a history of previous vascular surgery of involved limb
* Those who received hyperbaric oxygen therapy
* Those with unrelated skin disease around the involved foot will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult diabetic foot ulcer patients visiting endocrine department of tertiary care hospitals of Balochsitan, Pakistan with or with out amputation.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Baseline characteristics of amputees vs non amputees | 10 months
  Explore the baseline demographic, clinical, and lab investigations profile of diabetic foot patients visiting tertiary care hospitals of Baluchistan, Pakistan
Predictors of amputation in diabetic foot ulcer patient | 10 months
  Analyze the risk factors of amputation in diabetic foot ulcer patient

SECONDARY OUTCOMES:
Antibiotic resistance level | 10 months
  Explore the resistance level to most common antibiotics in diabetic foot ulcer patients

CONTACTS AND LOCATIONS:
Overall Officials: Shairzaman Khan, FCPS, Study Director — Bolan Univeristy of Medical and Health Sciences Quetta, Pakistan; Taimoor Hussain, MBBS, Principal Investigator — Bolan Medical Complex Hospital Quetta Pakistan
Locations (1):
- Bolan Medical Complex Hospital Quetta, Pakistan, Quetta, Balochistan, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Investigators will decide in future on how and when to share the IPD.

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Zhang P, Lu J, Jing Y, Tang S, Zhu D, Bi Y. Global epidemiology of diabetic foot ulceration: a systematic review and meta-analysis dagger. Ann Med. 2017 Mar;49(2):106-116. doi: 10.1080/07853890.2016.1231932. Epub 2016 Nov 3. PMID 27585063
- [Background] Alexiadou K, Doupis J. Management of diabetic foot ulcers. Diabetes Ther. 2012 Nov;3(1):4. doi: 10.1007/s13300-012-0004-9. Epub 2012 Apr 20. PMID 22529027
- [Background] Boulton AJ, Vileikyte L, Ragnarson-Tennvall G, Apelqvist J. The global burden of diabetic foot disease. Lancet. 2005 Nov 12;366(9498):1719-24. doi: 10.1016/S0140-6736(05)67698-2. PMID 16291066
- [Background] McEwen LN, Ylitalo KR, Herman WH, Wrobel JS. Prevalence and risk factors for diabetes-related foot complications in Translating Research Into Action for Diabetes (TRIAD). J Diabetes Complications. 2013 Nov-Dec;27(6):588-92. doi: 10.1016/j.jdiacomp.2013.08.003. Epub 2013 Sep 10. PMID 24035357
- [Background] Gershater MA, Londahl M, Nyberg P, Larsson J, Thorne J, Eneroth M, Apelqvist J. Complexity of factors related to outcome of neuropathic and neuroischaemic/ischaemic diabetic foot ulcers: a cohort study. Diabetologia. 2009 Mar;52(3):398-407. doi: 10.1007/s00125-008-1226-2. Epub 2008 Nov 27. PMID 19037626
- [Background] Yazdanpanah L, Shahbazian H, Nazari I, Arti HR, Ahmadi F, Mohammadianinejad SE, Cheraghian B, Hesam S. Incidence and Risk Factors of Diabetic Foot Ulcer: A Population-Based Diabetic Foot Cohort (ADFC Study)-Two-Year Follow-Up Study. Int J Endocrinol. 2018 Mar 15;2018:7631659. doi: 10.1155/2018/7631659. eCollection 2018. PMID 29736169
- [Background] Al-Rubeaan K, Al Derwish M, Ouizi S, Youssef AM, Subhani SN, Ibrahim HM, Alamri BN. Diabetic foot complications and their risk factors from a large retrospective cohort study. PLoS One. 2015 May 6;10(5):e0124446. doi: 10.1371/journal.pone.0124446. eCollection 2015. PMID 25946144